CLINICAL TRIAL: NCT01539148
Title: A Quality of Life Study Using Insulin Potentiation Targeted LowDose (IPTLDSM ) Chemotherapy and Nutrition Therapy in the Treatment of Cancer - The IPTLDSM QoL Broad Study
Brief Title: A Five-Year Quality of Life Study for Cancer Patients
Acronym: IPTLD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Constantine A. Kotsanis (Industry)
Collaborators: Best Answer for Cancer Foundation (Other)
Responsible Party: Sponsor-Investigator, Constantine A. Kotsanis, Principle Investigator, M.D., The Kotsanis Institute
Organization: The Kotsanis Institute (Industry)
Other Study IDs: 10.03.0010
Record Dates: First submitted 2012-02-16; First posted 2012-02-27 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Cancer
Keywords: Quality of Life; Qol; Questionnaire; Survey; Insulin Potentiation Targeted Low Dose Chemotherapy; IPTLD; Nutritional Therapy; Chemotherapy; Cancer Treatment; Kotsanis Institute; The Best Answer for Cancer Foundation; Liberty IRB; Texas
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigator is looking for patients who have been diagnosed with stage 1-4 cancer to enroll in a five year Quality of Life clinical trial study in which the participant has previously elected to use Insulin Potentiation Targeted Low Dose (IPTLD) as a means to treat their illness. This study is a quality of life study and not a treatment study. Participants participating in the study will be asked to complete quality of life questionnaires. The questionnaires completed by the patients will measure mood, energy level, ability to function, level of pain, and other measures that indicate how a patient feels about the quality of their daily living.

DETAILED DESCRIPTION:
Patients will complete surveys once per month during their participation in the quality of life study, and then a series of follow-up surveys: every two months the second year; every three (3) months the third year and every six months the fourth and fifth year.

ELIGIBILITY:
Inclusion Criteria:

* Only patients in active treatment with IPTLD are eligible i.e. patients have consented to treatment with IPTLD.
* Women who are pregnant, or could become pregnant, may not participate in the study.
* Patients 18 years of age or older
* Patients have to be able and willing to complete the various QoL instruments, which will be given upon enrollment and at designated follow-up intervals.
* Patients must have either had the benefits of standard, appropriate therapy and have had that fail, or refuse to receive these therapies after having been informed of the standard of care for their particular stage and diagnosis. This criteria is included for ethical, not clinical reasons.
* In addition, other criteria may be developed that more specifically address: The type, stage, location of the cancer/metastasis. The length of time since diagnosis. Previous treatments attempted and their outcome, Length of time since last treatment and concurrent conventional treatments. Nutritional approaches, other cam treatments, factors that may confound the study results.
* Ability, commitment of patient to follow IPTLD protocol
* Best Answer for Cancer Foundation and Kotsanis Institute do intend to draw subjects only from within the pool of patients who have elected to undergo IPTLD and nutrition therapy as their treatment of choice; limiting the universe of subjects to IPTLD patients removes the confounding effects of patient treatment choice and possible consideration of other treatment arms from the design.
* The focus is simple: it is to follow IPTLD patients and determine longitudinal impacts of treatment on quality of life experienced by IPTLD patients as a treatment group.
* It is to allow comparison with well-documented QoL results from conventional chemotherapy. This is the original intent, and recruitment efforts for participants will remain within those who are IPTLD patients.
* The initial, baseline QoL testing of IPTLD patients who choose to be in the study will include some questions designed to elicit the reasons the patient decided on IPTLD and nutrition therapy. Documenting these choices can serve two purposes; correlations between reasons, and the attitudes they reveal about factors known to impact QoL, such a positive sense of controlling one's health choices, can be drawn. Further, once these factors are accounted for, some inferences about the extent to which IPTLD and nutrition therapy are responsible for impacts on QoL can be derived.

Exclusion Criteria:

* The Medical Director/Principal Investigator will consider excluding specific cancers, for ethical reasons, that are intractable and known to have a rapid course, or which are known to be unresponsive to IPTLD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be from patients who have been diagnosed with stage 1-4 cancer that have chosen to use IPTLD and nutritional therapy and have been referred by a physician, word of mouth or through internet website inquiries.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Study | yearly
  MDASI Survey, FACIT

CONTACTS AND LOCATIONS:
Overall Officials: Constantine A. Kotsanis, MD, Principal Investigator — The Kotsanis Institute
Locations (1):
- The Kotsanis Institute, Grapevine, Texas, United States

REFERENCES:
- See also: The Kotsanis Institute — http://kotsanisinstitute.com